CLINICAL TRIAL: NCT04527289
Title: Potential Impact of Amantadine on Traumatic Brain Injury Outcomes
Brief Title: Impact of Amantadine on Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Amantadine on TBI
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Trauma, Brain
Keywords: traumatic brain injury (TBI); Interleukin-18 (IL-18); Neuron specific enolase (NSE); Neurotensin (NT)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Amantadine

STUDY DESIGN:
Intervention Model Description: All enrolled 50 patients will be divided into two groups; Group I are patients who will receive amantadine as add on therapy. Group II are patients who will be managed with the standard regimen.
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amantadine Group (Experimental): Group, I are patients who will receive amantadine (100mg) as add on therapy to the standard regimen.
  Interventions: Drug: Amantadine (100mg) as add on therapy.
- Placebo Group (Placebo Comparator): Group II are patients who will be managed with the standard regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine (100mg) as add on therapy. — Amantadine (100mg) as add on therapy to the management regimen of traumatic brain injury - 100mg twice daily Oral or feeding tube
  Other Names: PK-merz
  Arms: Amantadine Group
Drug: Placebo — patients will be managed with placebo as add on to the standard regimen.
  Arms: Placebo Group

SUMMARY:
The aim of this study is to evaluate whether the addition of amantadine to the management regimen of traumatic brain injury patients would have a favorable effect on recovery and neurological complications in association with prognosis biomarkers Interleukin-18 (IL-18), Neuron-specific enolase (NSE) and (Neurotensin).

DETAILED DESCRIPTION:
Proposal Steps

1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. All participants agreed to take part in this clinical study and provide informed consent.
3. Patients will be enrolled if they present with clinical signs of trauma, from Emergency department at Tanta University Hospital
4. Complete physical, laboratory, radiological assessment will be done for all patients
5. Serum samples will be collected for measuring the biomarkers.
6. All enrolled 50 patients will be divided into two groups; Group I are patients who will receive amantadine as added on therapy. Group II are patients who will be managed with the standard regimen.
7. All patients will be followed up during 6 weeks period.
8. At the end of 6 weeks, prognosis biomarkers will be withdrawn.
9. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
10. Measuring outcome: The primary outcome is to compare the effect of adding amantadine on recovery rate and neurological complications in trauma patients.
11. Results, conclusion, discussion and recommendations will be given.

Methodology

* 50 Patients will be randomized equally to the assigned study groups
* Prognosis biomarkers (IL-18, NSE and Neurotensin) will be measured using ELISA
* Conventional routine tests (including renal function tests) will be assessed
* Patients will be evaluated clinically (such as Glasgow score…) for recovery rate for neurological complications.

ELIGIBILITY:
* Inclusion criteria

  •Adult patients will be enrolled if they present with clinical signs of trauma brain injury
* Exclusion criteria

  * Age lower than 18
  * Females with positive pregnancy test
  * Known congestive heart failure or ischemic heart disease
  * Any injury disturbs the examination (high cervical cord injury or locked-in syndrome, could be a source of bias)
  * Penetrating head trauma
  * Need for any operation (laparotomy or craniotomy)
  * Severe brain disease (For example CVA history or brain tumour)
  * Renal failure with GFR lower than 60 ml/min
  * Patients with unknown identity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Neurotensin pg/ml | 2 weeks
  Neurotensin pg/ml by ELISA Kit
Neuron specific enolase (NSE) ng/mL | 2 Weeks
  Neuron specific enolase (NSE) by ELISA Kit
interleukin-18 (IL-18) pg/ml | 2 Weeks
  interleukin-18 (IL-18) by ELISA Kit
ICU stay (days) | 6 weeks
  ICU stay (days)

SECONDARY OUTCOMES:
(GCS) Total Glasgow Coma Scale score: (Severe: GCS 8 or less- Moderate: GCS 9-12- Mild: GCS 13-15). | 6 weeks
  number of GCS to describe the level of consciousness in a person following a traumatic brain injury.
GCS-E | 6 months
  The Glasgow Outcome Scale-Extended (GOS-E)

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Lecturer, Study Director — Damanhour University
Locations (1):
- Tanta University Hospital, Tanta, Elgarbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stelmaschuk S, Will MC, Meyers T. Amantadine to Treat Cognitive Dysfunction in Moderate to Severe Traumatic Brain Injury. J Trauma Nurs. 2015 Jul-Aug;22(4):194-203; quiz E1-2. doi: 10.1097/JTN.0000000000000138. PMID 26165872
- [Background] Bharosay A, Bharosay VV, Varma M, Saxena K, Sodani A, Saxena R. Correlation of Brain Biomarker Neuron Specific Enolase (NSE) with Degree of Disability and Neurological Worsening in Cerebrovascular Stroke. Indian J Clin Biochem. 2012 Apr;27(2):186-90. doi: 10.1007/s12291-011-0172-9. Epub 2011 Nov 8. PMID 23542317
- [Background] Ciaramella A, Della Vedova C, Salani F, Viganotti M, D'Ippolito M, Caltagirone C, Formisano R, Sabatini U, Bossu P. Increased levels of serum IL-18 are associated with the long-term outcome of severe traumatic brain injury. Neuroimmunomodulation. 2014;21(1):8-12. doi: 10.1159/000354764. Epub 2013 Sep 26. PMID 24080899